CLINICAL TRIAL: NCT03077971
Title: Effectiveness of Acceptance and Commitment Therapy Self-Help for Carers of People With Multiple Sclerosis: A Feasibility Randomised Controlled Trial
Brief Title: Effectiveness of Acceptance and Commitment Therapy Self-Help for Carers of People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: G14112016
Record Dates: First submitted 2017-02-28; First posted 2017-03-13 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Carer Stress Syndrome
Keywords: Carers of People with Multiple Sclerosis; Carer Strain; Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT Self-Help (Experimental): Participants in this arm will receive a self-help book based on Acceptance and Commitment Therapy (ACT). Participants will receive chapters each week, either electronically or by post, for 8 weeks.
  Interventions: Behavioral: ACT Self-Help
- ACT Self-Help with Telephone Support (Experimental): Participants in this arm will receive a self-help book based on Acceptance and Commitment Therapy (ACT). Participants will receive chapters each week, either electronically or by post, for 8 weeks. In addition to this, participants will have weekly telephone calls to support the use of the book.
  Interventions: Behavioral: ACT Self-Help with Telephone Support
- Treatment As Usual (No Intervention): Participants in this arm will have no intervention as part of the trial.

INTERVENTIONS:
Behavioral: ACT Self-Help — Self-Help Intervention Workbook using an Acceptance and Commitment Therapy approach
  Arms: ACT Self-Help
Behavioral: ACT Self-Help with Telephone Support — Self-Help Intervention Workbook using an Acceptance and Commitment Therapy approach alongside weekly telephone support calls
  Arms: ACT Self-Help with Telephone Support

SUMMARY:
This is a feasibility study to evaluate whether it is possible to conduct a larger study to evaluate whether providing psychological support to carers of people with MS is effective in reducing carer strain. Whilst not all carers experience distress as a result of their caring duties, some do. This study is testing the use of Acceptance and Commitment Therapy (ACT) in a self-help format. Participants will learn about and use ACT by reading a book provided to them by the study. One group will receive the ACT book, another will receive the same book alongside weekly telephone support to use the book, and a third group will act as a control group and therefore will not have extra support. Participants are allocated to the groups based on chance (a computer will decide group allocation). Participants will complete questionnaires before group allocation, and then again 3 months after they were allocated to a group, and one final time 6 months after group allocation. Those who receive the self-help book will get sent chapters each week for 8 weeks. The groups will be compared on scores from the questionnaires and complete feedback interviews with a subgroup of those who receive the book, to gain feedback about their experiences of the study.

ELIGIBILITY:
Inclusion Criteria:

* primary carer for a person with MS,
* English speaking (intervention and assessments are in English),
* able to give informed consent.
* score at least 21 on the Zarit Burden Interview (demonstrating a minimum of mild distress)

Exclusion Criteria:

* diagnosis of MS themselves
* psychiatric diagnosis
* inability to commit to the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
ZBI | 3 months
  Zarit Burden Interview as a measure of carer strain

SECONDARY OUTCOMES:
ZBI | 6 months
  Zarit Burden Interview as a measure of carer strain
MCSI | 3 months, 6 months
  Modified Carer Strain Index as a measure of carer strain
CAREQOL-MS | 3 months, 6 months
  CAREQOL- MS is a health-related quality of life scale designed for carers of people with MS
AAQ-II | 3 months, 6 months
  The Acceptance and Action Questionnaire is a measure of experiential avoidance and psychological inflexibility, consistent with the ACT model
CompACT | 3 months, 6 months
  The Comprehensive Assessment of Acceptance and Commitment Therapy measures important processes of ACT
Service Use Questionnaire | 3 months, 6 months
  The service use questionnaire will measure the frequency in which participants access health and social care services

OTHER OUTCOMES:
Feedback Interviews | 3 months
  A selection of those in the two intervention groups will be invited to complete an interview to give feedback about the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Roshan dasNair, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potter KJ, Golijana-Moghaddam N, Evangelou N, Mhizha-Murira JR, das Nair R. Self-help Acceptance and Commitment Therapy for Carers of People with Multiple Sclerosis: A Feasibility Randomised Controlled Trial. J Clin Psychol Med Settings. 2021 Jun;28(2):279-294. doi: 10.1007/s10880-020-09711-x. PMID 32144616